CLINICAL TRIAL: NCT07307079
Title: Effectiveness of Non-Invasive High-Frequency Oscillatory Ventilation vs Conventional Ventilation for Preterm Neonates With Respiratory Distress Syndrome Following Nasal CPAP Failure.
Brief Title: Non-Invasive High-Frequency Oscillatory Ventilation vs Conventional Ventilation for Preterm Neonates.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR-FARHAN-INDUS-HOSPITAL
Record Dates: First submitted 2025-12-02; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Invasive High-Frequency Oscillatory Ventilation Group (Experimental): Neonates were managed using a high-frequency oscillatory ventilator with a noninvasive nasal interface. Ventilator settings were adjusted to a mean airway pressure (MAP) of 8-12 cmH₂O, a frequency of 10 Hz, an amplitude adjusted to maintain optimal chest vibration, and an FiO₂ titrated to maintain SpO₂ between 90-94%.
  Interventions: Procedure: Non-Invasive High-Frequency Oscillatory Ventilation
- Conventional Ventilation Group (Experimental): Neonates received invasive ventilation through an endotracheal tube. Settings were adjusted to an initial tidal volume of 4-6 mL/kg, positive end-expiratory pressure (PEEP) of 4-6 cmH₂O, a respiratory rate of 30-50 breaths per minute, and FiO₂ titrated to maintain SpO₂ between 90-94%.
  Interventions: Procedure: Conventional Mechanical Ventilation

INTERVENTIONS:
Procedure: Non-Invasive High-Frequency Oscillatory Ventilation — Neonates were managed using a high-frequency oscillatory ventilator with a noninvasive nasal interface. Ventilator settings were adjusted to a mean airway pressure (MAP) of 8-12 cmH₂O, a frequency of 10 Hz, an amplitude adjusted to maintain optimal chest vibration, and an FiO₂ titrated to maintain SpO₂ between 90-94%.
  Arms: Non-Invasive High-Frequency Oscillatory Ventilation Group
Procedure: Conventional Mechanical Ventilation — Neonates received invasive ventilation through an endotracheal tube. Settings were adjusted to an initial tidal volume of 4-6 mL/kg, positive end-expiratory pressure (PEEP) of 4-6 cmH₂O, a respiratory rate of 30-50 breaths per minute, and FiO₂ titrated to maintain SpO₂ between 90-94%.
  Arms: Conventional Ventilation Group

SUMMARY:
Given the high burden of respiratory distress syndrome (RDS) and its complications in resource-constrained settings, identifying effective, low-risk interventions is imperative. The study aimed to assess the improvement in oxygenation and ventilation parameters initiating non-invasive high-frequency oscillatory ventilation (nHFOV) or conventional mechanical ventilation (CMV) and to compare the incidence of air leaks, sepsis, bronchopulmonary dysplasia (BPD), intraventricular hemorrhage (IVH), prolonged hospital stays, and short-term survival rates.

DETAILED DESCRIPTION:
Global neonatal care is moving toward lung-protective ventilation strategies to improve outcomes for preterm neonates. Evaluating the role of nHFOV in low- and middle-income countries (LMICs) like Pakistan not only helps address local healthcare challenges but also contributes to global efforts to optimize neonatal care across diverse settings. To best of my knowledge no such type of study has been conducted in Pakistan. This study is non-invasive and cost effective. The findings of this study could inform policy decisions and resource allocation in NICUs across Pakistan and other middle-income countries (LMICs).

ELIGIBILITY:
Inclusion Criteria:

* Neonates of any gender
* Gestational age between 26 and 36 weeks
* Diagnosed with RDS.
* Failed to respond to nCPAP treatment

Exclusion Criteria:

* Major congenital anomalies like congenital diaphragmatic hernia, dysmorphism and congenital heart diseases
* Early onset sepsis at the time of enrollment

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Improvement in ventilation parameter | 24 hours
  Improvement in ventilation parameter, measured by arterial blood gas analysis of the assigned ventilation modality was noted.

SECONDARY OUTCOMES:
Bronchopulmonary dysplasia | 36 weeks post-menstrual age
  Bronchopulmonary dysplasia was considered 'yes' if the patient required supplemental oxygen (>21% FiO₂) for ≥28 days to maintain oxygen saturation between 90-94%.
Sepsis | 28 days
  At least 1 abnormality in laboratory findings of WBC <5,000/mm³, I/T ratio >0.2, and platelets <100,000/mm³. or CRP elevated (>10 mg/L), or procalcitonin elevated (>2 ng/mL). or blood gas analysis metabolic acidosis (pH <7.25) was taken as 'yes'.
Ventilator-Associated Pneumonia | 48 hours
  Clinically, pneumonia was labeled 'yes' as a new or persistent respiratory distress or worsening gas exchange, increased ventilator requirements (e.g., higher FiO₂ or positive end-expiratory pressure [PEEP]), signs of infection (fever (>38°C) or hypothermia (<36°C), apnea or bradycardia episodes, tachycardia or hypotension).
Duration of respiratory support | 28 days
  Total days on modality were noted.
Survival Status at Discharge | 28 days
  The survival status of the patient was noted as 'alive' or 'deceased'.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Farhan, FCPS, Principal Investigator — Indus Hospital - Recep Tayyip Erdogan Campus, Muzaffargarh; Athar Razzaq, FCPS, Study Director — Indus Hospital - Recep Tayyip Erdogan Campus, Muzaffargarh
Locations (1):
- Indus Hospital - Recep Tayyip Erdogan Campus, Muzaffargarh, Muzaffargarh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.